CLINICAL TRIAL: NCT03610191
Title: Serum Biomarkers for Prediction and Diagnosis of POCD in Elderly Patients Undergoing Cardiac Surgery.
Brief Title: MD2, Cystatin C and DNA Methylation Tags as Serum Biomarkers for POCD.
Acronym: BM-POCD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, Lize Xiong, Professor, Xijing Hospital
Other Study IDs: KY20182029-1
Record Dates: First submitted 2018-07-03; First posted 2018-08-01 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Postoperative Cognitive Dysfunction
Keywords: biomarkers; MD2; Cystatin C; DNA methylation markers; SNP mutations in CTNNA2 gene
MeSH Terms: conditions — Postoperative Cognitive Complications | interventions — Cardiac Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient serum with DNA fragments
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgery: Patients aged over 18 scheduled for elective cardiac surgery under CPB and general anesthesia. This group will later be divided in to two sub groups based on their neuropsychological battery tests results before surgery and one day before discharge. Blood sample will be collected before, immediately after surgery and at 24h after surgery for serum biomarker tests: MD2, CysC as well as DNA methylation markers of neural system origin.
  Interventions: Diagnostic Test: Serum biomarker tests; Behavioral: Neuropsychological battery tests; Procedure: Cardiac surgery
- non-surgical control: Age and sex matched volunteers from the community were included for neuropsychological battery tests and set as controls for the diagnosis of POCd in surgical patients.
  Interventions: Behavioral: Neuropsychological battery tests

INTERVENTIONS:
Diagnostic Test: Serum biomarker tests — Blood was collected at preoperatively, immediately after operation and 24 h after operation in patients from the surgical group but not volunteers. Serum MD2, CysC, DNA methylation marker and SNP mutation sites on CTNNA2 gene were test.
  Groups: Surgery
Behavioral: Neuropsychological battery tests — both surgical patients and volunteers will accept three times of NPB tests. For surgical patients the tested time point are preoperative, one day before discharge and 3 months after surgery. For volunteers the tested time interval would be similar to that of surgical patients.
  Other Names: NPB tests
Procedure: Cardiac surgery — patients scheduled for cardiac surgery will accept the surgical procedure.
  Groups: Surgery

SUMMARY:
Postoperative cognitive dysfunction (POCD) is a severe complication after surgery. Currently, a complicated battery of neuropsychological tests both before and after surgery with other characteristics-matched population as control are needed for the diagnosis of POCD. This diagnosis is also delayed, which could not be used to screen for high risk patients who may need intervention beforehand. The current trial targeted a surgical population of elderly patients undergoing cardiac surgery under cardiopulmonary bypass (CPB), which is a population of the highest incidence of POCD, to screen for possible predictive or diagnostic biomarkers in the serum for POCD. Myeloid differentiation factor 2 (MD2), also known as lymphocyte antigen 96, is a protein involved in biding lipopolysaccharide with Toll like receptor-4 (TLR4). Recently the investigators have found that increased MD2 expression in the hippocampus of the mice after surgery stimuli. On the other hand, the investigators have reported that cystatin C (CysC) as an endogenous neuroprotective factor for stroke. It may also be involved in endogenous neural protection against POCD. This trial is to investigate whether serum MD2, CysC can be used for prediction and diagnosis of POCD in surgical population. Serum based DNA methylation biomarkers will also be tested for prediction or diagnosis of POCD development. Also in our orevious research, SNPs cites at rs6739405、rs12467815、rs12472215、rs11126727、rs11126731、rs993607 were revealed as possible susceptibility variations for POCD (diagnosed with MMSE only, NCT02084030) in patients undergoing CPB. This study will also test the SNP variations in study populations to varify if one or conbination of morethan one of these varuations can be a risk factor for POCD when diagonosed with NPT.

DETAILED DESCRIPTION:
Postoperative cognitive dysfunction (POCD) is a common complication of surgical patients, which manifested by reduced memory, attention and calculation abilities etc. Among different types of surgeries, the incidence of POCD in cardiac surgical patients are the highest, the prevalence of POCD on the day of discharge was as high as 53%, and 26% of patients still showed cognitive dysfunction three months after surgery. POCD can increase patients' hospitalization days, increase the consumption of medical resources and social security resources, seriously affect patients' postoperative quality of life, and even increase the mortality rate one year after surgery. There is no definite serum marker for the prediction and diagnosis of POCD. The diagnosis currently applied are a series of neuropsychological battery tests both before and after surgery. it's both time consuming and inapplicable to patients in severe conditions. The purpose of this trial is to screen out POCD serum markers as effective indicators for POCD prediction, early diagnosis of POCD, and assessment for therapeutic efficacy.

At present, the pathogenesis of POCD is not clear. Aging, general anesthesia, heart surgery, preoperative cognitive impairment and cardiovascular diseases are high risk factors for POCD. At present, preoperative and postoperative neuropsychological behavior assessments is the only way to diagnose POCD, but it is time consuming, resource occupying, and also has learning effect. However, studies on serum markers that can predict the risk of POCD or for early diagnosis of POCD are still at a very preliminary stage. Study has found that plasma inflammatory factors: interleukin (IL)-1β, IL-8 and tumor necrosis factor-α level raised in POCD patients [1-2]. In addition, in microglial cells, inflammatory reaction mediated by S100β modulated the receptor for advanced glycation end products (RAGE) signaling pathway [3], and raise pro-inflammatory factor expressions [4], so S100β expression may be related to POCD occurrence. However, inflammatory related factors such as IL-1, IL-8 and TNF-α lack neurological or disease specificity. S100B, previously thought to have diagnostic effects of nerve injury, has not been confirmed in small sample correlation studies [5]. Therefore, it is of great clinical significance to collect reliable and powerful clinical research data to explore serum biomarkers for early prediction and diagnosis of POCD.

The investigators have previously found that higher endogenous CystatinC level is an important protective mechanism against ischemic brain injury. Elevated serum Cystatin C, accompanied with brain cystatin C level elevation, can inhibit lysosome damage, promote autophagy [6] and induce ischemic tolerance in the brain. Myeloid differentiation protein (MD-2) is a secreted protein, composed of 160 amino acids and participate in TLR4 signaling pathway, mediated inflammatory response [7]. The investigator using an animal model of POCD also found that the MD2 expression is significantly increased after surgery.

In addition, the methylation is an important modification way of proteins and nucleic acids, it regulates the expression of genes and is closely related to many diseases such as alzheimer's. Studies have shown that COASY and SPINT1[17], NCAPH2/LMF2[18] promoter region DNA methylation has diagnostic value for alzheimer's disease and mild cognitive impairment. Therefore, we speculate that changes in the DNA methylation markers of the central nervous system may be of early diagnostic value for POCD after cardiac surgery. Therefore, the detection of the central nervous system methylation label in the serum of patients after cardiac surgery will provide a new research direction for the clinical detection of central nervous system injury.

Our previous clinical trial (NCT 02084030) indicates that, 6 SNP mutations on the CTNNA2 gene (SNPs cites at rs6739405、rs12467815、rs12472215、rs11126727、rs11126731、rs993607) has altered risk for POCD in elderly patients undergoing CPB. Since this gene functions as a linker between cadherin adhesion receptors and the cytoskeleton to regulate cell-cell adhesion and differentiation in the nervous system, it also regulates morphological plasticity of synapses and cerebellar and hippocampal lamination during development, we aim to verify if patients that has any of these mutations is more susceptible to POCD then patients that has none, or less of these mutations, using a more integrated neuropsychological test battery tests as compared to MMSE used in the previous trial.

In conclusion, the investigators believe that serum central nerveous system (CNS) specific methylation markers, MD2 level and CystatinC level may have predictive and diagnostic value for POCD. This trial is to to evaluate POCD in 200 patients with cardiac surgery under CPB, test their perioperative serum MD2, CystatinC, and DNA methylation markers from the central nervous system, and explore their role in prediction and diagnosis of POCD.

ELIGIBILITY:
Inclusion Criteria:

* Patients age≥18 yrs scheduled for coronary artery bypass graft (CABG), valve replacement or CABG+valve replacement surgery under CPB and general anesthesia in Xijing Hospital, from Nov, 2018.

Exclusion Criteria:

* Has neurodegenerative disease: dementia, Alzheimer's or Parkinson's Disease
* Has received neuropsychological tests before
* Psychological disorder that needs medication
* Preoperative Mini-Mental State Examination (MMSE)< 24
* Didn't finish elementary school
* Has symptomatic cerebrovascular disease.
* Has received cardiac surgery or neurosurgery before
* Has cardiac arrest experience and received cardiopulmonary resuscitation
* Renal dysfunction (serum creatinine>2 mg/dL or 176.82 μmol/L)
* Hepatic pathology (AST, ALT exceeded 1.5 times of the upper limit of normal range)
* Unable to comply or non-cooperative
* Can't finish process under instruction
* Can't understand mandarin
* Has severe visual or auditorial impairment
* Has severe alcohol or drug dependence (has been drinking over 100 ml of ≥50° alcohol per day , for over 3 months. And other drug abuse problem)
* Has been enrolled in the same study before or is currently involved in other clinical trials.

Ages: 18 Years to 108 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery under cardio-pulmonary bypass (CPB) and general anesthesia. Non-surgical controls are age and gender-matched community residents.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2018-11-20 (Actual); Primary Completion 2021-09-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Preoperative serum MD2/CysC/DAN Methylation marker/SNPs mutation rates on CTNNA2 gene before anesthesia | Immediately before anesthesia
  Blood samples will be collected at immediately before anesthesia and tested for MD2/CysC/DAN Methylation marker value.
Postoperative serum MD2/CysC/DAN Methylation marker/immediately after surgery | Immediately after surgery
  Blood samples will be collected at immediately after surgery and tested for MD2/CysC/DAN Methylation marker value.
Postoperative serum MD2/CysC/DAN Methylation marker value at 24 h after surgery | Twenty-four hours after surgery
  Blood samples will be collected at 24h after surgery and tested for MD2/CysC/DAN Methylation marker value.
Neuropsychological battery (NPB) assessment | From one day before surgery to 3 months after surgery
  NPB will be evaluated at 3 time points: 1. one day before surgery. 2. one day before discharge. 3. 3 months after surgery. The NPB includes: 1. Grooved Pegboard Test; 2. Auditory Word Memory Test; 3. Trail Making Test (Part A, Part B); 4. Digit Span Test; 5. Digit Symbol Subtest; 6. Verbal Fluency Test; and 7. Word Recall Test.
  POCD at discharge or 3 months after surgery will be analyzed as follow: 2 or more tests of the NPB with a Z score over 1.96 or less than -1.96, patient is defined as POCD. And patients that have less than 2 tests with a Z score over 1.96 is defined as no-POCD.
  Note: the time frame of postoperative NPB test is defined as one day before discharge. It is usually within 5-9 days depending on the hospitalization time for each patient. Since NPB test is time consuming and requires patients at a comfortable state. The investigators chose one day before discharge as many clinical trials regarding POCD reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, M.D., Ph.D., Principal Investigator — Xijing Hospital, the Fourth Military Medical University
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Li YC, Xi CH, An YF, Dong WH, Zhou M. Perioperative inflammatory response and protein S-100beta concentrations - relationship with post-operative cognitive dysfunction in elderly patients. Acta Anaesthesiol Scand. 2012 May;56(5):595-600. doi: 10.1111/j.1399-6576.2011.02616.x. Epub 2012 Jan 9. PMID 22224444
- [Background] Bi Y, Liu S, Yu X, Wu M, Wang Y. Adaptive and regulatory mechanisms in aged rats with postoperative cognitive dysfunction. Neural Regen Res. 2014 Mar 1;9(5):534-9. doi: 10.4103/1673-5374.130084. PMID 25206851
- [Background] Bianchi R, Adami C, Giambanco I, Donato R. S100B binding to RAGE in microglia stimulates COX-2 expression. J Leukoc Biol. 2007 Jan;81(1):108-18. doi: 10.1189/jlb.0306198. Epub 2006 Oct 5. PMID 17023559
- [Background] Li RL, Zhang ZZ, Peng M, Wu Y, Zhang JJ, Wang CY, Wang YL. Postoperative impairment of cognitive function in old mice: a possible role for neuroinflammation mediated by HMGB1, S100B, and RAGE. J Surg Res. 2013 Dec;185(2):815-24. doi: 10.1016/j.jss.2013.06.043. Epub 2013 Jul 17. PMID 23899512
- [Background] Linstedt U, Meyer O, Kropp P, Berkau A, Tapp E, Zenz M. Serum concentration of S-100 protein in assessment of cognitive dysfunction after general anesthesia in different types of surgery. Acta Anaesthesiol Scand. 2002 Apr;46(4):384-9. doi: 10.1034/j.1399-6576.2002.460409.x. PMID 11952437
- [Background] Fang Z, Deng J, Wu Z, Dong B, Wang S, Chen X, Nie H, Dong H, Xiong L. Cystatin C Is a Crucial Endogenous Protective Determinant Against Stroke. Stroke. 2017 Feb;48(2):436-444. doi: 10.1161/STROKEAHA.116.014975. Epub 2016 Dec 20. PMID 27999137
- [Background] Kobayashi N, Shinagawa S, Nagata T, Shimada K, Shibata N, Ohnuma T, Kasanuki K, Arai H, Yamada H, Nakayama K, Kondo K. Usefulness of DNA Methylation Levels in COASY and SPINT1 Gene Promoter Regions as Biomarkers in Diagnosis of Alzheimer's Disease and Amnestic Mild Cognitive Impairment. PLoS One. 2016 Dec 19;11(12):e0168816. doi: 10.1371/journal.pone.0168816. eCollection 2016. PMID 27992572